CLINICAL TRIAL: NCT04937465
Title: CTR025 FAUN - Hydration Status
Brief Title: Explorative Study on a New Device' Ability to Register Hydration Change in Elderly Subjects During Rehabilitation.
Status: Withdrawn | Type: Observational
Why Stopped: Study was stopped because of covid-19 restrictions imposed for the next 9 months
Sponsor: Mode Sensors AS (Industry)
Collaborators: Norwegian Computing Center, Oslo Norway (Unknown); Lilleborg helsehus, Oslo, Norway (Unknown); Nidarvoll helsehus, Trondheim, Norway (Unknown); Ryen helsehus, Trondheim, Norway (Unknown); Solvang helsehus, Oslo, Norway (Unknown); Søbstad helsehus, Trondheim, Norway (Unknown); Øya helsehus, Trondheim, Norway (Unknown)
Responsible Party: Sponsor
Other Study IDs: CTR002 FAUN
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-06

CONDITIONS: Dehydrated, Water-Electrolyte Imbalance, Malnutrition
MeSH Terms: conditions — Dehydration; Water-Electrolyte Imbalance; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples: osmolality, hemoglobin, platelets, leukocytes, sodium, glucose potassium, creatinine, Glomerular filtration rate (GFR), albumin, calcium,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly: Elderly (> 70 yrs) eligible for a short term rehabilitation
  Interventions: Other: No intervention done

INTERVENTIONS:
Other: No intervention done — No intervention was done. This was an observational study.

SUMMARY:
Test the ability of continuous measurements from a new sensor patch to set the hydration state in subjects who are malnourished/dehydrated or overhydrated or otherwise not optimally hydrated. Specifically, clinical examination, blood pressure, blood tests, and weight change at the admission and at the discharge will be used to establish the true hydration status of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients eligible for rehabilitation

Exclusion Criteria:

* Subjects with end stage cancer

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly people eligible for short term (3 - 5 weeks) rehabilitation because of either (i) malnutrition and or dehydration, or (ii) overhydration from heart failure treatment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Hydration state | During rehabilitation period (3 - 5 weeks)
  Set correct hydration state with a sensitivity of 0.90 and a specificity of 0.80

CONTACTS AND LOCATIONS:
Locations (6):
- Norway (6):
  - Lilleborg helsehus, Oslo
  - Ryen helsehus, Oslo
  - Solvang helsehus, Oslo
  - Øya helsehus, Trondheim
  - Nidarvoll helsehus, Trondheim
  - Søbstad helsehus, Trondheim

IPD SHARING:
Plan to Share IPD: No